CLINICAL TRIAL: NCT05865093
Title: Early Visual Functions in Patients at Risk of Developing Cerebral Visual Impairment. A Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Ricci Daniela, Principal Investigator Pediatric Neurologist, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5006
Record Dates: First submitted 2023-03-17; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess visual function from neonatal age to 36 months of age in infants at risk of visual impairment due to brain lesion or ocular pathology

ELIGIBILITY:
Inclusion Criteria:

* Age between 34 weeks of post-menstrual age and 36 months of life in children born before 37 weeks gestational age
* Genetic syndroms
* Hypoxic Hischemic Encephalopathy
* Brain malformation
* Metabolic diseases
* Ocular pathologies

Exclusion Criteria:

* Patients at low risk of developing neurological outcomes
* Refusal of informed consent

Ages: 2 Days to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children at risk for visual impairment due to brain lesion, brain malformation, genetic syndroms, Hypoxic Hischemic Encephalopathy, metabolic diseases or ocular pathologies, assessed at neonatal age and followed up to 36 months of age
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Early Visual Functions in Patients at Risk of Developing Cerebral Visual Impairment. A Pilot Study | 5 years
  The score of the functional visual assessment will be obtained at neonatal age and at 1-3-6-9-12-18-24-36 months of life will be analysed at each age and compared to neurodevelopment findings using different scales according to age.
  These results will be related to the MRI total score (obtained by the sum of scores by site: cortex, basal ganglia, white matter and cerebellum, normal (0), mild abnormal (1), severely abnormal (2)).

SECONDARY OUTCOMES:
Correlation betwwen functional visual assessment score to MRI score | 5 years
  Results of functional visual assessment will be related to the MRI total score (obtained by the sum of scores by site: cortex, basal ganglia, white matter and cerebellum, normal (0), mild abnormal (1), severely abnormal (2)).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy